CLINICAL TRIAL: NCT02430480
Title: Neoadjuvant Androgen Deprivation and Enzalutamide: Using Multiparametric MRI to Evaluate Intraprostatic Tumor Responses and Androgen Resistance Patterns in Newly Diagnosed Prostate Cancer
Brief Title: Using Multiparametric MRI to Evaluate Intraprostatic Tumor Responses and Androgen Resistance Patterns in Newly Diagnosed Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Fatima Karzai, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 150124; 15-C-0124
Record Dates: First submitted 2015-04-28; First posted 2015-04-30 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Multiparametric MRI; Prostatectomy; Focal Prostate Cancer; Normal Testosterone; Non-Metastatic
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Goserelin; enzalutamide; Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 1/Arm 1- Enzalutamide and Goserelin (Experimental): Patients will have an multi-parametric magnetic resonance imaging (mpMRI) guided biopsy, then receive enzalutamide and goserelin subcutaneous (SC) treatment for 6 months followed by a second mpMRI examination.
  Interventions: Drug: Goserelin; Drug: Enzalutamide; Device: mpMRI

INTERVENTIONS:
Drug: Goserelin — 10.8mg administered subcutaneously every 12 weeks (2 doses)
  Other Names: Zoladex
Drug: Enzalutamide — 160mg orally, daily for 24 weeks
  Other Names: ASP-9785
Device: mpMRI — Multiparametric MRI - One at baseline and after 6 months of treatment
  Other Names: multi-parametric magnetic resonance imaging

SUMMARY:
Background:

* There are several ways to treat prostate cancer. Researchers want to see how well a certain kind of imaging helps detect prostate cancer. They also want to see if a particular drug combination used before surgery will benefit people with prostate cancer that hasn't spread in the body (non-metastatic). The combination will be androgen deprivation therapy and enzalutamide.
* The combination of androgen deprivation therapy and enzalutamide has been shown to make patients with advanced (metastatic disease) live longer. The investigators want to see if using it earlier can increase cure rate of surgery and identify genetic or molecular characteristics that are associated with better outcomes.

Objectives:

- To develop better ways of detecting prostate cancer before and after pre-operative treatment.

Eligibility:

- Men at least 18 years old with non-metastatic prostate cancer. They must be candidates for a radical prostatectomy.

Design:

* Participants will be screened with medical history, physical exam, and blood tests. They will have scans and X-rays.
* Before starting the study drugs, participants will have:
* Vital signs taken, medical history, and blood tests.
* Electrocardiogram (ECG) heart test, with patches stuck on the skin.
* Small piece of tumor removed (biopsy) using image guidance from magnetic resonance imaging (MRI) and ultrasound.
* 3T multi-parametric magnetic resonance imaging (mpMRI). Participants will lie on a table that slides into a metal cylinder. A probe will be inserted in the rectum. They will be in the scanner for about 60 minutes, lying still. The scanner makes loud knocking sounds. Participants will get earplugs.
* Participants will take the 2 study drugs for 6 months.
* Enzalutamide is taken as 4 pills once a day.
* Androgen deprivation therapy is given by injection 2 times over 6 months.
* During these 6 months, participants will visit the clinic monthly. They will have physical exam, vital signs, and blood drawn.
* After finishing the study drugs, participants will have another 3T mpMRI. Then they will have prostate removal surgery.

DETAILED DESCRIPTION:
Background:

* Most men diagnosed with prostate cancer will present with intermediate or high-risk disease
* Many develop castrate resistant prostate cancer (CRPC) as curative strategies are often unsuccessful
* Treatment options typically involve radical prostatectomy (RP) or radiation therapy (RT) in combination with androgen deprivation therapy (ADT)
* Even when cancers are initially sensitive to ADT, resistance ultimately emerges either through clonal selection or through a variety of adaptive mechanisms (secondary resistance).
* The recent introduction of novel androgen pathway inhibitors offers an opportunity to potentially improve the cure rate of men with intermediate and high risk localized prostate cancer
* There remains a great need for improved techniques to determine mechanisms of treatment response and resistance.

Objectives:

-To test the feasibility of multi parametric magnetic resonance imaging (mpMRI) for the localization and detection of focal prostate cancer both before and after pre-operative treatment with ADT and enzalutamide.

Eligibility:

* Patients with nonmetastatic castration sensitive prostate cancer with intermediate or high-risk features
* Patients with testosterone levels greater than or equal to 100 ng/dL.
* Eastern Cooperative Oncology Group (ECOG) 0-1.

Design:

* Patients will be treated with ADT and enzalutamide for 6 months
* Two 3T mpMRI endorectal examinations (One at screening and after 6 month of treatment)
* Screening biopsy (magnetic resonance (MR)/ultrasound (US) guided) samples
* Standard of care prostatectomy (RP) following post treatment mpMRI
* All tumor specimens will undergo genomic analysis

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed prostate cancer confirmed by the Laboratory of Pathology, National Cancer Institute (NCI) or Pathology Department at Walter Reed Bethesda
* Must have previously untreated (with definitive therapy) prostate cancer with intermediate or high risk features defined as:

  * Intermediate risk:

    * Prostate-specific antigen, (PSA) level is between 10 and 20 ng/ml or
    * Gleason score is 7 or
    * Stage T2b or T2c
  * High Risk:

    * Gleason 8 and higher OR
    * PSA greater than 20 at the time of diagnosis OR
    * Seminal vesicle involvement OR
    * Possible (on magnetic resonance imaging (MRI) Extra-capsular extension (T3 disease)
* Patients must be eligible for and must be planning to undergo radical prostatectomy
* Patients must have testosterone levels greater than or equal to 100 ng/dL
* Men age greater than or equal to 18 years.

  * Children are excluded because prostate cancer is not common in pediatric populations.
  * Women are not eligible because this disease occurs only in men.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1
* Patients must have normal organ and marrow function as defined below:
* Hemoglobin greater than or equal to 9 g/dL
* leukocytes greater than or equal to 3,000/mcL
* absolute neutrophil count greater than or equal to 1,500/mcL
* platelets greater than or equal to 150,000/mcL
* total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST)/Serum glutamic-oxaloacetic transaminase(SGOT)/Alanine aminotransferase (ALT) Serum glutamic pyruvic transaminase (SGPT) less than or equal to 3 X institutional upper limit of normal
* creatinine within normal institutional limits

OR

* creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
* The effects of enzalutamide on the developing human fetus are unknown. For this reason and because androgen receptor antagonists as well as other therapeutic agents used in this trial are known to be teratogenic, male participants and their female partners of child bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence). Male participants should use a condom if having intercourse with a pregnant woman. Additionally, a condom plus another effective method of birth control is recommended during therapy and for 3 months after treatment for male participants having intercourse with a woman of reproductive potential. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Willingness to undergo biopsy.
* Ability to detect lesions within prostate on magnetic resonance imaging (MRI) for biopsy
* Willingness to travel to National Institutes of Health (NIH) for follow-up visits.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents (in the past 28 days) or herbal medications (within 1 day).
* Patients with distant metastatic disease beyond N1(regional) lymph nodes on conventional imaging studies (Computed tomography (CT), MRI or Bone Scan).
* Patients who have received any prior therapy for prostate cancer with surgery, radiation, and/or chemotherapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to enzalutamide or other agents used in study.
* Clinically significant cardiac disease, e.g. New York Heart Association (NYHA) classes III-IV; uncontrolled angina, uncontrolled arrhythmia or uncontrolled hypertension, myocardial infarction in the previous 6 months as confirmed by an electrocardiogram (ECG).
* Contraindication to biopsy:

  * Bleeding disorders
  * Prothrombin Time (PT)/Partial Thromboplastin Time (PTT) greater than or equal to 1.5 times the upper limit of normal
  * Artificial heart valve
* Contraindication to MRI:

  * Patients weighing more than weight limit for the scanner tables
  * Allergy to MR contrast agent
  * Patients with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic device
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with known human immunodeficiency virus (HIV) are eligible. These patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. In addition, if patients are receiving combination antiretroviral therapy, there is potential for pharmacokinetic interactions with enzalutamide. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients with known active treatment for Hepatitis B and C infections.
* Patients who are taking medications that are strong inhibitors of Cytochrome P450 3A4 (CYP3A4) or P-glycoprotein (PgP) and need to remain on these medications. For a current table of Substrates, Inhibitors and Inducers please access the following website:

http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm

* History of seizure, including any febrile seizure, loss of consciousness, or transient ischemic attack, or any condition that may pre-dispose to seizure (e.g., prior stroke, brain arteriovenous malformation, head trauma with loss of consciousness requiring hospitalization).
* Other medications used for urinary symptoms including 5-alpha reductase inhibitors (finasteride and dutasteride) and alternative medications known to alter prostate specific antigen (PSA) (eg phytoestrogens and saw palmetto) cannot be taken while patients are receiving enzalutamide
* Patients with a malignancy within the past 3 years for which study drugs or a prostatectomy is a contraindication.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Karzai, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to the Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Wilkinson S, Ku AT, Lis RT, King IM, Low D, Trostel SY, Bright JR, Terrigino NT, Baj A, Summerbell ER, Heyward KE, Kartal S, Fenimore JM, Li C, Singler C, Vo B, Jansen CS, Ye H, Whitlock NC, Harmon SA, Carrabba NV, Atway R, Lake R, Takeda DY, Kissick HT, Pinto PA, Choyke PL, Turkbey B, Dahut WL, Karzai F, Sowalsky AG. Localized high-risk prostate cancer harbors an androgen receptor activity-low subpopulation susceptible to HER2 inhibition. J Clin Invest. 2025 Sep 4;135(22):e189900. doi: 10.1172/JCI189900. eCollection 2025 Nov 17. PMID 40906535
- [Derived] Rathi N, Blake Z, Hyman J, Nemirovsky DR, Gelikman DG, Hesswani C, Koller C, Nethala D, Mendhiratta N, Kenigsberg AP, Noun J, Dahut W, Karzai FY, Linehan WM, Pinto PA, Turkbey B, Gurram S. Castration Levels of Testosterone Results in Atrophy of Androgen-sensitive Perineal Muscles: A Potential Biomarker for Male Hypogonadism. Urology. 2025 Feb;196:313-320. doi: 10.1016/j.urology.2024.10.006. Epub 2024 Oct 18. PMID 39427924
- [Derived] Karzai F, Walker SM, Wilkinson S, Madan RA, Shih JH, Merino MJ, Harmon SA, VanderWeele DJ, Cordes LM, Carrabba NV, Bright JR, Terrigino NT, Chun G, Bilusic M, Couvillon A, Hankin A, Williams MN, Lis RT, Ye H, Choyke PL, Gulley JL, Sowalsky AG, Turkbey B, Pinto PA, Dahut WL. Sequential Prostate Magnetic Resonance Imaging in Newly Diagnosed High-risk Prostate Cancer Treated with Neoadjuvant Enzalutamide is Predictive of Therapeutic Response. Clin Cancer Res. 2021 Jan 15;27(2):429-437. doi: 10.1158/1078-0432.CCR-20-2344. Epub 2020 Oct 6. PMID 33023952
- [Derived] Gold SA, VanderWeele DJ, Harmon S, Bloom JB, Karzai F, Hale GR, Marhamati S, Rayn KN, Mehralivand S, Merino MJ, Gulley JL, Bilusic M, Madan RA, Choyke PL, Turkbey B, Dahut W, Pinto PA. mpMRI preoperative staging in men treated with antiandrogen and androgen deprivation therapy before robotic prostatectomy. Urol Oncol. 2019 Jun;37(6):352.e25-352.e30. doi: 10.1016/j.urolonc.2019.01.012. Epub 2019 Apr 15. PMID 31000430
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0124.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
Started | 39
Completed | 36
Not Completed | 3
Not completed — Death | 1
Not completed — Anesthesia concerns | 1
Not completed — Progressed on treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 18
Age, Continuous [Median (Full Range); unit: years] | 61 [58 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 28
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 39
Median Prostate-Specific Antigen (PSA) at Baseline [Median (Full Range); unit: ng/ml] — Normal PSA is 0 to 4 ng/ml. Above 4ng/ml indicates cancer of the prostate.
  ng/ml | 9.56 [1.18 to 985.9]
Number of Participants Pre-Treatment Clinical Stage at Baseline [Count of Participants; unit: Participants] — Prostate Cancer Staging TNM system. T = tumor, N = nodes, M = metastasized.
  Stages of cancer is numbered from 1-4. A lower number (i.e. 1) means less cancer spread and a higher number (i.e. 4) means more cancer spread. Also, alphabetical letters a, b, and c can be used to denote lower or higher stages of the disease. A lower letter = lower stage of disease and a higher number = higher stage of disease.
  Participants
    T2 | 6
    T3a | 17
    T3b | 11
    T4 | 5
    N1 | 11
Median Prostate Volume on Magnetic Resonance Imaging at Baseline [Median (Full Range); unit: cc] — Prostate volume on magnetic resonance imaging (MRI) is calculated by 0.52 x length x width x height. Normal volume should be less than 25 cc's. Greater than 25 cc's is an enlarged prostate (bad) as it can cause symptoms (i.e.: nocturia, difficulty emptying, etc.)
  cc | 42.0 [33.0 to 49.0]
Median Prostate Specific Antigen (PSA) Density [Median (Full Range); unit: ng/ml^2] — PSA density is defined as a calculation performed at diagnosis and is the serum prostate specific antigen (PSA) level (ng/mL) divided by the volume of the prostate gland (mL).
  PSA density ≤0.08 is low risk for prostate cancer and ≥0.08 is high risk for prostate cancer.
  ng/ml^2 | 0.22 [0.15 to 0.39]
Median Magnetic Resonance Tumor Burden [Median (Full Range); unit: Ratio] — Relative tumor burden (RTB) volumes were calculated by dividing the combined volumes of each lesion divided by the prostate volume.
  Ratio | 3.47 [1.9 to 9.8]
Number of Participants in a Gleason Group (biopsy) [Count of Participants; unit: Participants] — There is a prostate cancer grading system, called the Grade Groups with groups 1 through 5 based on how much cancer cells look like normal prostate tissue under the microscope. If the cancerous tissue looks much like normal prostate tissue, a grade of 1 is assigned. If the cancer cells and their growth patterns look very abnormal, a grade of 5 is assigned. Grades 2 through 4 have features in between these extremes. The higher the grade, the more likely it is that the cancer will grow and spread quickly.
  Participants
    1 | 0
    2 | 6
    3 | 5
    4 | 11
    5 | 17
Number of Participants in a Risk-Group [Count of Participants; unit: Participants] — Gleason score is calculated by adding the score of the most common grade (Gr) (primary Gr pattern) and the 2nd most common Gr (secondary Gr pattern) and ranges from 6-10. The individual primary and secondary Gr patterns range from 1-5. Higher Gleason scores = a higher Gr of prostate cancer, i.e., a more advanced or more aggressive type of cancer. Per protocol Intermediate risk is PSA10 and 20ng/ml or Gleason score 7 or Stage T2b (i.e. cancer in about 3/4 of the prostate) or T2c (i.e. cancer in entire prostate). High risk is Gleason score ≥8 or PSA>20 at dx or seminal vesicle involvement.
  Participants
    Intermediate | 3
    High | 36

OUTCOME MEASURES:

1. Primary Outcome: Median Tumor Volume Burden at Baseline Multi-parametric Magnetic Resonance Imaging (mpMRI) Before and After Surgery
Description: The prostate lesion is contoured manually by an expert radiologist. Research software (mim-vista) calculates the volume. Greater tumor volumes may indicate higher prostate tumor growth.
Time Frame: Baseline and 6 months
Population: 37 out of 39 patients completed treatment and underwent pre- and post- mpMRI. Two patients did not-one patient died on study from a recreational drug overdose. The other had progression of disease on study.
Measure: Median (Full Range); unit: cc
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
Number analyzed (Participants) | 37
cc
  Baseline | 3.44 [0.44 to 54.75]
  6 months | 0.62 [0 to 102.4]

2. Secondary Outcome: Median Nuclear Androgen Receptor (AR) Level in Biopsy Specimens Versus Residual Tumors
Description: The effect of intense androgen suppression and inhibition was measured on tumors using anti-AR immunostains of biopsy and surgical specimens. Detection of tumor nuclear AR was quantified on a per-nucleus basis using computer-aided image analysis with Definiens Developer XD 64, grouping nuclei into high, medium, low, and absent bins, a histology score was assigned to each sample.
  Nucleus classification is low vs. med. at 0.7; med. vs. high at 0.95. Definiens reported the total # of positively stained nuclei or cells, along with the distribution of low-, med.-, and high-intensity stained nuclei/cells for ea. tumor focus. A %positive index score was calculated using a weighted avg. divided by the total # of objects, where index = [ (1 × nuclei/cells stained low) + (2 × nuclei/cells stained med.) + (3 × nuclei/cells stained high) ](3 × total nuclei).
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
Number analyzed (Participants) | 37
scores on a scale
  biopsy specimen | 0.7568 [-0.5 to 0.87]
  residual tumor | 0.1661 [0 to 0.7]

3. Secondary Outcome: Median Prostate Lesion Volume Before and After Treatment
Description: Prostate lesion volumes on baseline and post-treatment multiparametric magnetic resonance imaging (mpMRI) were calculated from T2W-MRI sequences using software embedded in the PACS after manual contouring by the same radiologist. Lesion volume scores were categorized as low (2 or fewer positive sequences), moderate (3 positive sequences) and high (4 positive sequences). Lesion volume values are in cubic centimeters (cc's).
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: cubic centimeters
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
Number analyzed (Participants) | 37
cubic centimeters
  Baseline | 39.5 [18.9 to 73]
  6 months | 20.0 [10.1 to 103]

4. Secondary Outcome: Number of Participants With a Complete Response
Description: Complete response was evaluated after neoadjuvant treatment with androgen deprivation therapy (ADT) and enzalutamide and assessed by pathologic exam. Pathologic complete response: the absence of residual invasive cancer confirmed by immunohistochemistry (IHC).
Time Frame: After neoadjuvant treatment with androgen deprivation therapy (ADT) and enzalutamide, approximately 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
Number analyzed (Participants) | 37
Participants | 2

5. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 51 months and 2 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
Number analyzed (Participants) | 39
Participants | 38

6. Secondary Outcome: Number of Prostate Lesions Detected Within the Study Population at Baseline Multi-parametric Magnetic Resonance Imaging (mpMRI) and 6 Months After Enzalutamide Plus Androgen Deprivation Therapy (ADT)
Description: Prostate lesion volumes on baseline and post-treatment mpMRI were calculated from T2W-MRI sequences using software embedded in the PACS after manual contouring by the same radiologist.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Number; unit: Lesions
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
Number analyzed (Participants) | 37
Lesions
  Baseline | 58
  6 months | 40

7. Secondary Outcome: Initial Multiparametric Magnetic Resonance Imaging (mpMRI) Percentage of Relative Tumor Volume Sensitivity
Description: The Youden index was used as a measure for evaluating biomarker effectiveness and was calculated to determine the cutoffs that gave the optimal combination of sensitivity and speciﬁcity for patient response to treatment. The index is: J=sensitivity + specificity -1. Its value ranges from 0 through 1 (inclusive). A value of 1 indicates that there are no false positives or false negatives, i.e. the test is perfect. The index gives equal weight to false positive and false negative values, so all tests with the same value of the index give the same proportion of total misclassified results. Sensitivity and specificity are the probability of truly identifying relative tumor burden on multiparametric magnetic resonance imaging (mpMRI) respectively at a statistically established cut point.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: Percentage of sensitivity
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
Number analyzed (Participants) | 37
Percentage of sensitivity | 81

8. Secondary Outcome: Number of Participants With Reduction in Phosphatase and Tensin Homolog (PTEN) Levels
Description: PTEN level reduction was evaluated using immunohistochemistry in post treatment specimens. For anti-PTEN immunohistochemistry, a case was considered PTEN-reduced (abnormal) if at least 5% of tumor cells demonstrated reduced PTEN intensity relative to PTEN in benign cells (lower than 5%, then abnormal).
Time Frame: post treatment, approximately 1-3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
Number analyzed (Participants) | 37
Participants | 21

9. Secondary Outcome: Number of Participants With Positive Erythroblast Transformation-specific (ETS)-Related Gene (ERG) Protein Overexpression
Description: ERG protein overexpression was evaluated using immunohistochemistry in post treatment specimens. A positive ETS-related ERG overexpression is a bad outcome.
Time Frame: Approximately one month-3 months post-treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
Number analyzed (Participants) | 37
Participants | 14

10. Secondary Outcome: Initial Multiparametric Magnetic Resonance Imaging (mpMRI) Percentage of Relative Tumor Volume Specificity
Description: as for outcome 7
Time Frame: 6 months
Measure: Number; unit: Percentage of specificity
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
Number analyzed (Participants) | 36
Percentage of specificity | 87

11. Other Pre Specified Outcome: Any Grade 1 Adverse Events in More Than One Patient and Grades 2 -3 Attributable to Research
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event (i.e., Grade 1) is any untoward medical occurrence. A serious adverse event (i.e., Grade 2-3) is an adverse event or suspected adverse reaction that results in an adverse drug experience, and/or disruption of the ability to conduct normal life functions attributable to the research.
Time Frame: Date treatment consent signed to date off study, approximately 51 months and 2 days.
Measure: Number; unit: Adverse events
Groups:
- Grade 1: Common Terminology Criteria for Adverse Events (CTCAE) v4
  Grade 1 is Mild; asymptomatic or mild symptoms.
- Grade 2: Common Terminology Criteria for Adverse Events (CTCAE) v4 Grade 2 is moderate, minimal.
- Grade 3: Common Terminology Criteria for Adverse Events (CTCAE) v4 Grade 3 is severe or medically significant but not immediately life threatening,
Arm/Group | Grade 1 | Grade 2 | Grade 3
Number analyzed (Participants) | 39 | 39 | 39
Adverse events
  Fatigue | 20 | 2 | 0
  Edema, limbs | 2 | 0 | 0
  Erectile dysfunction | 9 | 3 | 1
  Gynecomastia | 3 | 0 | 0
  Hot flashes | 34 | 1 | 0
  Hypertension | 1 | 7 | 7
  Confusion | 2 | 0 | 0
  Libido decreased | 15 | 0 | 0
  Insomnia | 12 | 4 | 0
  Mood changes | 2 | 0 | 0
  Personality change | 3 | 0 | 0
  Restlessness | 2 | 1 | 0
  Headache | 5 | 0 | 0
  Dizziness | 5 | 0 | 0
  Memory impairment | 3 | 0 | 0
  Concentration impairment | 3 | 0 | 0
  Dysuria | 1 | 1 | 0
  Urinary incontinence | 2 | 4 | 0
  Dysgeusia | 1 | 1 | 0
  Dyspepsia | 2 | 0 | 0
  Nausea | 4 | 0 | 0
  Cough | 3 | 0 | 0
  Sore throat | 2 | 0 | 0
  Arthralgia | 2 | 0 | 0
  Back pain | 3 | 0 | 0
  Muscle weakness | 2 | 0 | 0
  Myalgia | 2 | 1 | 0
  Rash | 1 | 2 | 0
  Weight gain | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 51 months and 2 days.
Arm/Group | 1/Arm 1- Enzalutamide and Goserelin
All-Cause Mortality (participants affected / at risk) | 1/39
Serious Adverse Events (participants affected / at risk) | 2/39
Other Adverse Events (participants affected / at risk) | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Arm 1- Enzalutamide and Goserelin (N=39)
Sudden death NOS (General disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Arm 1- Enzalutamide and Goserelin (N=39)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bladder spasm (Renal and urinary disorders) | 2 (2)
Blurred vision (Eye disorders) | 3 (3)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Cholesterol high (Investigations) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 3 (3)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 3 (3)
Ejaculation disorder (Reproductive system and breast disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 12 (12)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Fatigue (General disorders) | 23 (24)
Fever (General disorders) | 1 (1)
Floaters (Eye disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Diverticulitis with symptoms of anorexia, abd pain and nausea with retching but no vomiting
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Gynecomastia (Reproductive system and breast disorders) | 3 (3)
Headache (Nervous system disorders) | 6 (6)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hot flashes (Vascular disorders) | 35 (36)
Hypertension (Vascular disorders) | 17 (28)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) — Blunt force trauma
Insomnia (Psychiatric disorders) | 15 (16)
Libido decreased (Psychiatric disorders) | 15 (15)
Lymphocele (Vascular disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Otitis media (Ear and labyrinth disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 4 (4)
Perineal pain (Reproductive system and breast disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Personality change (Psychiatric disorders) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Prostatic pain (Reproductive system and breast disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Psychiatric disorders - Other, Mood changes (Psychiatric disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (6)
Renal calculi (Renal and urinary disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 6 (6)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 7 (9)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 10 (10)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (4)
Urinary urgency (Renal and urinary disorders) | 5 (7)
Ventricular arrhythmia (Cardiac disorders) | 3 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Weight gain (Investigations) | 2 (4)
Weight loss (Investigations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT02430480/Prot_SAP_004.pdf
  • Informed Consent Form (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT02430480/ICF_003.pdf